CLINICAL TRIAL: NCT02101437
Title: The Relationship of Platelet Micro-RNA Expression and Platelet Reactivity in Patients Under Clopidogrel or Ticagrelor Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Yueh-Chung, Chen, chief of ICU, Taipei City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TCHIRB-I021003
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2017-04

CONDITIONS: PRU; miRNA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- control (Placebo Comparator): normal subjects.
  Interventions: Procedure: miRNA within 24hr; Procedure: miRNA after 1 week; Procedure: miRNA after 1 month
- clopidogrel (Active Comparator): subjects received clopidogrel 75mg qd.
  Interventions: Procedure: miRNA within 24hr; Procedure: miRNA after 1 week; Procedure: miRNA after 1 month
- ticagrelor (Active Comparator): subjects received ticagrelor 90mg qd.
  Interventions: Procedure: miRNA within 24hr; Procedure: miRNA after 1 week; Procedure: miRNA after 1 month
- cilostazol (Active Comparator): subjects received cilostazol 100mg bid.
  Interventions: Procedure: miRNA within 24hr; Procedure: miRNA after 1 week; Procedure: miRNA after 1 month

INTERVENTIONS:
Procedure: miRNA within 24hr — miRNA within 24hr
Procedure: miRNA after 1 week — miRNA after 1 week
Procedure: miRNA after 1 month — miRNA after 1 month

SUMMARY:
For acute coronary syndrome patients undergoing cardiac catheterization after stenting, we will give dual antiplatelet drugs (dual antiplatelet agents) therapy, the choice of the basis of medical criteria (clinical guidelines) routine as aspirin + clopidogrel or aspirin + ticagrelor, according to medical guidelines currently no other disposal alternative proposal (unless adverse drug tolerance or bleeding can not be administered); idea of this experiment for acute coronary syndrome or conventional cardiac catheterization after stenting, platelet miRNA expression (miR-96 , miR-200b, miR-495, miR-107) after cardiac catheterization and interventional treatment of clopidogrel or ticagrelor acceptance of platelet reactivity (PRU) correlation values (given clopidogrel or ticagrelor determined by the clinician, the patient follow-up experiment to track only and observation), aims to explore under different platelet reactivity (hyper-reactive or hypo-reactive), their differences in miRNA performance.

ELIGIBILITY:
Inclusion Criteria:

1 under DAPT (dual antiplatelet therapy) of stable angina patients for elective stent implantation.

2. DAPT 24 hours after treatment PRU (platelet activity units) values. (Drug unresponsive patients was defined as PRU> 235).

Exclusion Criteria:

1.Not suitable for the treatment of patients with DAPT. (Active peptic ulceration or bleeding) 2 patients of aspirin, clopidogrel, ticagrelor, cilostazol medication intolerance.

3 contraindications for aspirin, clopidogrel, ticagrelor, cilostazol drug usage (such as heart failure patients not suitable for use cilostazol).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: chen yueh chung, chieft, Principal Investigator — taipei city hospital cardiovascular section
Locations (1):
- Taipei city hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen YC, Lin FY, Lin YW, Cheng SM, Chang CC, Lin RH, Chuang CL, Sheu JS, Chen SM, Tsai CS. Platelet MicroRNA 365-3p Expression Correlates with High On-treatment Platelet Reactivity in Coronary Artery Disease Patients. Cardiovasc Drugs Ther. 2019 Apr;33(2):129-137. doi: 10.1007/s10557-019-06855-3. PMID 30783954

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: no stent or anti-platelet drugs
- Clopidogrel: under clopidogrel treatment
- Ticagrelor: under ticagrelor treatment
- Clopidogrel+Cilostazol: under clopidogrel and cilostazol treatment
Period: Overall Study
Arm/Group | Control | Clopidogrel | Ticagrelor | Clopidogrel+Cilostazol
Started | 20 | 54 | 52 | 49
Completed | 20 | 54 | 52 | 49
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: receive different anti-platelet drugs
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Clopidogrel | Ticagrelor | Clopidogrel+Cilostazol | Total
Number analyzed (Participants) | 20 | 54 | 52 | 49 | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 12 | 12 | 56
  >=65 years | 6 | 36 | 40 | 37 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.67 (9.81) | 66.39 (10.68) | 67.99 (13.56) | 65.35 (11.55) | 66.59 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 14 | 21 | 59
  Male | 12 | 38 | 38 | 28 | 116
Region of Enrollment [Number; unit: participants]
  Taiwan | 20 | 52 | 54 | 49 | 175

OUTCOME MEASURES:

1. Primary Outcome: miRNA
Description: miRNA-365-3p measure by Roche miRNA kits; PRP(platelet riched plasma) isolated miRNA by isolation Kit, then havest in cDNA synthesis Kit; then perform RT PCR.
  .
Time Frame: 7 days
Population: check miRNA expression: Normalized expression level=2 -Ct, which means the more amount of miRNA, the less Ct.
  Negative valure indicated expression<1, and calculated after log2; the final was fold change expression of miRNA-365-3p compared to the control sample.
Measure: Mean (Full Range); unit: fold of change
Arm/Group | Control | Clopidogrel | Ticagrelor | Clopidogrel+Cilostazol
Number analyzed (Participants) | 20 | 54 | 52 | 49
fold of change | -8.14 [-8.48 to -7.61] | -3.46 [-5.1 to -0.63] | -7.54 [-8.27 to -6.81] | -3.97 [-5.26 to -3.62]

ADVERSE EVENTS:
Arm/Group | Control | Clopidogrel | Ticagrelor | Clopidogrel+Cilostazol
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/54 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/54 | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 0/20 | 0/54 | 0/52 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No